CLINICAL TRIAL: NCT03355963
Title: Comparative Study Between Intracavernosal Injection of Botulinum Toxin Type A (50 and 100 Unit) Efficacy and Durability in the Treatment of Vascular Erectile Dysfunction
Brief Title: Intracavernosal Injection of Botulinum Toxin Type A (50 and 100 Unit) in the Treatment of Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-Shaer, MD, Principal Investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-09-2016
Record Dates: First submitted 2017-11-13; First posted 2017-11-29 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Erectile Dysfunction; Botulinum Toxin
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sodium Chloride; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Placebo Comparator): The control group: received an IC 1 ml saline injection one day after the penile Doppler/trimix test.
  Interventions: Other: saline injection
- Group B (Active Comparator): The treatment group B: received a single IC injection of BTX-A 50 units one day after the penile Doppler/trimix test.
  Interventions: Biological: Botulinum toxin type A 50 units
- Group C (Active Comparator): The treatment group C:
  intervention: received a single IC injection of BTX-A 100 units one day after the penile Doppler/trimix test.
  Interventions: Biological: Botulinum toxin type A 100 units

INTERVENTIONS:
Other: saline injection — The control group: received an IC 1 ml saline injection one day after the penile Doppler/trimix test.
  Other Names: group A (control group)
  Arms: Group A
Biological: Botulinum toxin type A 50 units — The treatment group B: received a single IC injection of BTX-A 50 units one day after the penile Doppler/trimix test.
  Other Names: group B
  Arms: Group B
Biological: Botulinum toxin type A 100 units — The treatment group C: received a single IC injection of BTX-A 100 units one day after the penile Doppler/trimix test.
  Other Names: group C
  Arms: Group C

SUMMARY:
purpose: The aim of this study is to compare the safety, efficacy and durability of different doses of BTX-A (50 and 100 unit) in the treatment of Vasculogenic Erectile Dysfunction after failure of other ICI therapy.

Patients and Methods: This study will be conducted on 200 patients diagnosed as vascular erectile dysfunction by penile color Doppler not responding to medical and injection therapy presenting to Urology department and outpatient clinic at Benha University Hospital, Andrology, Sexology & STD's outpatient clinic, Kasr El Aini Hospitals, Cairo University.(multicentric study).

A- Inclusion criteria:

* Age between 40 to 70 years.
* Vascular ED proved by penile duplex.
* Unable to develop erections sufficient for intercourse.
* A "No" response on Sexual encounter profile questions (SEP 2 & 3)
* Failing to respond to first line and second line treatments for Erectile Dysfunction with surgery as the only remaining treatment option.

B-Exclusion criteria:

* Significant cardiovascular disease interfering with sexual activity
* Any history of an unstable medical or psychiatric condition
* Any presence of penile anatomical abnormalities (e.g. penile fibrosis) that would significantly impair erectile function.

patients will be simply randomized into 3 equal groups, one control group and two treatment groups. Ethics committee approval and informed consent were obtained.

DETAILED DESCRIPTION:
introduction: Evidence has been arising suggesting that Botulinum toxin type A (BTX-A) injections can relax smooth muscles fibers in the treatment of obesity and Detrusor muscle over-activity, similar effect on cavernosal smooth muscles would help in the treatment of erectile dysfunction (ED) resistant to oral and intracavernous (IC) therapy, thus avoiding surgical treatment options.

patient and methods: All patients will perform penile color Doppler evaluation to confirm a vascular etiology, a trimix solution (PGE1 10 ug + Phentolamine 1 mg + Papaverine 30 mg) was injected IC during the penile Doppler study.

The control group: received an IC 1 ml saline injection one day after the penile Doppler/trimix test.

The treatment group B: received a single IC injection of BTX-A 50 units one day after the penile Doppler/trimix test.

The treatment group C: received a single IC injection of BTX-A 100 units one day after the penile Doppler/trimix test.

Assessment for all groups was done by penile color Doppler exam, Sexual Health Inventory for men (SHIM), Sexual Encounter Profile questions 2 and 3 (SEP 2 & SEP 3), and the global assessment question (GAQ) were completed pre-treatment and 2 weeks after treatment also, 3 and 6 months after treatment.

Procedure:

At least 1 day after the penile color Doppler test, the patient is placed in the supine position flaccid and stretched penile length and girth would be measured from tip of the penis to the pubic bone will be done. A rubber band will be applied to the base of the penis. The skin will be prepped with alcohol swabs followed by the IC injection of 50 units of BTX-A for patients in treatment group B and 100 units of BTX-A for patients in treatment group C with direct pressure will be applied for 2 minutes. The rubber band will be removed after 15 minutes.

Patients and controls will fill the Sexual Health Inventory for men (SHIM) questionnaire and answer the ,Sexual Encounter Profile questions 2 and 3 (SEP 2 & SEP 3), and the global assessment question (GAQ) before and 2 weeks, 3 months and 6 months after treatment .

The rational for selecting the minimum 2-weeks waiting period is to give a chance for the BTX-A to reach its maximum effect. Possible Risks include pain and prolonged erections, also 3 months and 6 months after treatment do detect safety, efficacy and durability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 to 70 years. Vascular ED proved by penile duplex. Unable to develop erections sufficient for intercourse. A "No" response on Sexual encounter profile questions (SEP 2 & 3) Failing to respond to first line and second line treatments for Erectile Dysfunction with surgery as the only remaining treatment option.

Exclusion Criteria:

* Significant cardiovascular disease interfering with sexual activity Any history of an unstable medical or psychiatric condition Any presence of penile anatomical abnormalities (e.g. penile fibrosis) that would significantly impair erectile function.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Erectile Function (EF) domain score of the International Index of Erectile Function (IIEF) | pre-treatment and 2 weeks after treatment also, 3 and 6 months after treatment
  Changes in the Erectile Function (EF) domain score of the International Index of Erectile Function (IIEF) between treatment periods and baseline in different study arms. the score as follow:
  > 7 severe dysfunction 7-12 Moderate dysfunction
  13-18 Mild to moderate dysfunction
  19-24 Mild dysfunction
  25-30 No dysfunction
the Sexual Event Profile (SEP) scores | baseline, 2 weeks post treatment , 3, and 6 months post treatment
  Changes in the Sexual Event Profile (SEP) scores between treatment periods and baseline in different study arms by a <yes or no> response .
Global Assessment Questionnaire (GAQ) scores | baseline, 2 weeks post treatment , 3, and 6 months post treatment
  Changes in the Global Assessment Questionnaire (GAQ) scores between treatment periods in different study arms by a <yes or no> response
Cavernosal artery peak systolic and end diastolic velocities | baseline, 2 weeks post treatment , 3, and 6 months post treatment
  Change in Peak systolic velocity in the Cavernosal arteries, on color Doppler examination, in the patient and control groups.